CLINICAL TRIAL: NCT07347223
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of DD-S052P in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of DD-S052P in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HLB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DD-S052P-P1
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: DD-S052P; Phase 1; First-in-Human; Healthy Volunteers; Single Ascending Dose; Intravenous Administration; Safety; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive either DD-S052P or placebo in parallel cohorts within single ascending dose and multiple ascending dose parts.
Who Masked: Care Provider
Masking Description: Participants, investigators, care providers, and outcome assessors are blinded to treatment assignment. Study drug and placebo are identical in appearance and administered in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DD-S052P (SAD/MAD) (Experimental): Participants receive DD-S052P administered as an intravenous infusion over 4 hours. Single ascending doses (SAD) or multiple ascending doses (MAD) are evaluated to assess safety, tolerability, and pharmacokinetics in healthy volunteers.
  Interventions: Drug: DD-S052P
- Placebo (SAD/MAD) (Placebo Comparator): Participants receive placebo (Ringer solution) administered as an intravenous infusion over 4 hours, matching the dosing schedule of the DD-S052P treatment in the single and multiple ascending dose cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DD-S052P — DD-S052P is administered as an intravenous infusion at single or multiple ascending dose levels to evaluate safety, tolerability, and pharmacokinetics in healthy adult subjects.
  Arms: DD-S052P (SAD/MAD)
Drug: Placebo — Placebo solution administered as an intravenous infusion, matching the investigational product in appearance, volume, and administration schedule.
  Arms: Placebo (SAD/MAD)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, first-in-human study designed to evaluate the safety, tolerability, and pharmacokinetics of DD-S052P in healthy adult volunteers.

The study consists of two parts: a single ascending dose (SAD) part and a multiple ascending dose (MAD) part. In the SAD part, participants will receive a single intravenous infusion of DD-S052P or placebo at increasing dose levels. In the MAD part, participants will receive multiple intravenous infusions of DD-S052P or placebo over several days.

Safety and tolerability will be assessed through monitoring of adverse events, vital signs, physical examinations, electrocardiograms (ECGs), and clinical laboratory tests. Pharmacokinetic assessments will be performed to characterize plasma concentrations of DD-S052P over time following single and multiple dosing.

The results of this study will provide important information to support further clinical development of DD-S052P.

DETAILED DESCRIPTION:
This Phase 1 study is a randomized, double-blind, placebo-controlled, first-in-human clinical trial designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of DD-S052P following intravenous administration in healthy adult subjects.

The study consists of two sequential parts: a single ascending dose (SAD) part and a multiple ascending dose (MAD) part.

In the SAD part, cohorts of healthy subjects will receive a single intravenous infusion of DD-S052P or placebo at escalating dose levels. Dose escalation to the next cohort will occur only after a review of available safety and tolerability data from the preceding cohort, in accordance with predefined stopping and escalation criteria.

In the MAD part, healthy subjects will receive multiple intravenous doses of DD-S052P or placebo administered once daily over consecutive days. Dose levels for the MAD part will be selected based on the safety, tolerability, and pharmacokinetic results obtained from the SAD part.

Safety and tolerability will be evaluated throughout the study by monitoring adverse events (AEs) and serious adverse events (SAEs), vital signs, physical examination findings, electrocardiograms (ECGs), and clinical laboratory parameters.

Pharmacokinetic assessments will be conducted to characterize plasma concentration-time profiles of DD-S052P following single and multiple dosing. Key pharmacokinetic parameters will be derived using standard non-compartmental methods, as appropriate.

The results of this study will provide essential information on the safety profile and pharmacokinetic characteristics of DD-S052P and will support further clinical development.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male/female aged to 18-50 years inclusive at the screening visit
2. Must agree to adhere to the contraception requirements:

   1. Female must be of non-childbearing potential, defined as meeting at least one of the following:

      * hysteroscopic sterilization
      * bilateral tubal ligation or bilateral salpingectomy
      * hysterectomy
      * bilateral oophorectomy
      * be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
   2. Female of childbearing potential who are sexually active must agree to use at least one highly effective method of contraception starting from the 1 month prior to first administration of the study drug until 4 months post-dosing:

      * Hormonal methods: oral, transdermal, systemic, or implantable contraceptives
      * Intrauterine devices (IUDs)
      * Barrier methods: condoms or diaphragms used with spermicide
      * Surgical sterilization of the male partner
   3. Male must use of condom by the male subject plus an effective method of contraception for the subject partner of childbearing potential from study drug administration until 4 months post-dosing (oral, transdermal, systemic or implant contraception birth control, intrauterine devices, diaphragm, surgical sterilization, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle)
3. Male subjects must not donate sperm from the first dosing until 90 days after the last dosing
4. Non-smoker subject or smoker of not more than 5 cigarettes a day
5. Body Mass Index (BMI) between 18.5 and 32.0 (kg/m2) inclusive, with body weight between 60 and 100 kg inclusive, at Screening and Day -1
6. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination)
7. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 min in supine position:

   * 95 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg,
   * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
   * 50 bpm ≤ HR ≤ 90 bpm,
   * Or considered not clinically significant (NCS) by investigators;
8. Normal ECG recording on a 12-lead ECG at the screening visit:

   * 120 < PR < 210 ms,
   * QRS < 120 ms,
   * QTcF ≤ 430 ms for male and QTcF ≤ 450 ms for female
   * No sign of any trouble of sinusal automatism,
   * Or considered NCS by investigators
9. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non-relevant by the Investigator
10. Normal dietary habits
11. Signing a written informed consent prior to participation
12. Subject with estimated Glomerular Filtration Rate (eGFR) ≥ 80 mL/min/1.73 m2, as estimated using CKD-EPI creatinine Equation (2021)

Exclusion Criteria:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, infectious disease; endocrine, immunologic, dermatologic or/and any relevant disease
2. Subject with proteinuria, Grade 2 or higher (CTCAE, Ver.5.0)
3. Symptomatic hypotension whatever the decrease of the blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within 2 min of changing from supine to standing position
4. Positive urine drug testing or alcohol testing at Screening or Day -1
5. Positive Hepatitis B surface antigen (HBsAg) or anti-Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
6. Clinical symptoms suspected of acute infectious disease within 2 weeks before the first study drug administration
7. Any medication intake (except acetaminophen) within 1 month or within 5 times the elimination half-life of the medication (whichever is longer) prior to the first administration of study drug
8. Serious or severe adverse reaction, including hypersensitivity, anaphylaxis or hepatotoxicity to carbapenems, cephalosporins, penicillins, polyethylene glycol derivatives, monobactams or any other medication
9. History of hypersensitivity to Ringer solution
10. Blood donation (including as part of a clinical trial) within 2 months before administration
11. General anaesthesia within 3 months before administration
12. Inability to abstain from intense muscular effort
13. Subjects who cannot be reliably contacted in case of an emergency
14. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses/day)
15. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem or poor mental development
16. Persons deprived of their liberty by judicial or administrative decision; persons under coercive psychiatric care; adults under legal protection (guardianship/trusteeship); persons under court protection
17. Participation in any interventional study within 60 days or within 5 times the elimination half-life of the interventional study drug (whichever is longer) before study check-in
18. Pregnant or breastfeeding or intended to become pregnant during the study
19. Any other reasons identified by the investigator that would preclude the subject's participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first study drug administration through the end-of-study visit (approximately up to Day 8 for Part A [SAD] and up to Day 14 for Part B [MAD]).
  Safety and tolerability will be evaluated by summarizing the number of participants experiencing one or more treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) following administration of DD-S052P.
  Adverse events will be assessed by the Investigator for severity and relationship to study drug. Severity grading will follow CTCAE v5.0, where applicable.
Change From Baseline in Vital Signs | From baseline (pre-dose) through the end-of-study visit (approximately up to Day 8 for Part A [SAD] and up to Day 14 for Part B [MAD]).
  Change from baseline will be assessed for the following vital sign parameters:
  systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (beats per minute), oral body temperature (°C), oxygen saturation (SpO₂, %), and respiratory rate (breaths per minute).
Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters | From baseline (pre-dose) through the end-of-study visit (approximately up to Day 8 for Part A [SAD] and up to Day 14 for Part B [MAD]).
  Change from baseline will be assessed for the following 12-lead ECG parameters:
  QT interval corrected using Fridericia's formula (QTcF, ms), PR interval (ms), and QRS duration (ms).
Number of Participants With Clinically Significant Abnormal Laboratory Results | From baseline through the end-of-study visit (approximately up to Day 8 for Part A [SAD] and up to Day 14 for Part B [MAD]).
  Clinically significant abnormal laboratory findings will be summarized as the number of participants with one or more abnormal laboratory results, as assessed by the Investigator.
  Laboratory assessments include hematology, serum chemistry/biochemistry, coagulation parameters, thyroid function tests, and urinalysis.

CONTACTS AND LOCATIONS:
Locations (1):
- HLB Science, Seoul, Seoul, South Korea